CLINICAL TRIAL: NCT00204763
Title: Comparison of Solid-State Esophageal Manometry and Water Perfused Anorectal Manometry Catheters With Air Filled Multi-Balloon Esophageal and Anorectal Manometry Catheters
Brief Title: Comparison of Esophageal and Anorectal Manometry Catheters
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We determined that the results would not be worth reporting.
Sponsor: University of Utah (Other)
Collaborators: Clinical Innovations (Industry)
Responsible Party: University of Utah, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12127
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Achalasia; Nutcracker Esophagus; Scleroderma; Esophageal Spasm; Fecal Incontinence
Keywords: manometry catheters; diffuse esophageal spasm or hypertensive LES; incontinence
MeSH Terms: conditions — Esophageal Achalasia; Esophageal Motility Disorders; Scleroderma, Diffuse; Esophageal Spasm, Diffuse; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Solid state catheter
  Interventions: Device: Solid state catheter
- A (Experimental)
  Interventions: Device: Air filled balloon catheter

INTERVENTIONS:
Device: Air filled balloon catheter — The new air filled balloon catheter will be tested against the solid state catheter
  Other Names: Clinical innovations manometry catheter
  Arms: A
Device: Solid state catheter — The standardly used solid state catheter will be tested against the new air filled balloon catheter
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the accuracy of esophageal and anorectal manometric pressure measurements using a newly developed air filled balloon catheter with present standard solid state esophageal and anorectal catheters, respectively.

DETAILED DESCRIPTION:
Twenty subjects with abnormal esophageal motility (5 subjects each with achalasia, nutcracker esophagus, scleroderma, diffuse esophageal spasm or hypertensive LES) previously referred for clinical esophageal motility testing will be contacted. These twenty subjects must have previously undergone esophageal manometry testing using the standard clinical protocol at the University of Utah motility with solid state manometry catheters. After obtaining informed consent, these twenty subjects will undergo the esophageal manometry using air-filled balloon catheters per the standard clinical protocol. Following the repeat procedure a short one-page questionnaire will be completed by the subject and the motility nurse.

Five subjects with the diagnosis of incontinence previously referred for clinical anorectal motility testing will be contacted. These five subjects must have previously undergone anorectal manometry using the standard clinical protocol for an anorectal manometry study with water perfused anorectal manometry catheters. After obtaining informed consent, these five subjects will undergo the anorectal manometry using air-filled balloon catheters per the standard clinical protocol. Following the repeat procedure a short one-page questionnaire will be completed by the subject and the motility nurse.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80 years old
* Ability to give informed consent
* No significant medical conditions
* Abnormal esophageal motility
* Abnormal anorectal motility

Exclusion Criteria:

* Previous esophageal or anorectal surgery, anatomic abnormalities or dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To compare the accuracy of esophageal and anorectal manometric pressure measurements using a newly developed air filled balloon catheter with present standard solid state esophageal and anorectal catheters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John C Fang, M.D., Principal Investigator — University of Utah HSC
Locations (1):
- University of Utah HSC, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Fang JC, Hilden K, Tuteja AK, Peterson KA. Comparison of air-coupled balloon esophageal and anorectal manometry catheters with solid-state esophageal manometry and water-perfused anorectal manometry catheters. Dig Dis Sci. 2004 Oct;49(10):1657-63. doi: 10.1023/b:ddas.0000043382.59539.d3. PMID 15573923